CLINICAL TRIAL: NCT03954054
Title: Evaluation of a Therapeutic Education Programme for Harm Reduction in People With Alcohol Use Disorder
Brief Title: Therapeutic Education for Harm Reduction in People With Alcohol Use Disorder
Acronym: ETHER
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Regional Agency for Health PACA (Other); SESSTIM UMR1252 (Aix-Marseille Univ, INSERM, IRD) (Unknown)
Responsible Party: Sponsor
Other Study IDs: C19-03 / ETHER
Record Dates: First submitted 2019-05-09; First posted 2019-05-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2021-03

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol; substance use; patient education; psychosocial skills; controlled drinking; harm reduction; abstinence; quality of life
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Harm Reduction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Former therapeutic education participants: Semi-structured interviews with people who already completed the TPE programme
  Interventions: Behavioral: "Choizitaconso" - therapeutic patient education programme
- Intervention group (current therapeutic education participants): A face-to-face interview and a telephone interview at treatment initiation (M0) and 6 months after programme initiation (M6)
  Administration of socio-economic questionnaires and a Brief Evaluation of Alcohol-Related Neuropsychological Impairment (BEARNI) before, and 6 months after inclusion in the therapeutic education programme.
  Interventions: Behavioral: "Choizitaconso" - therapeutic patient education programme
- Control AUD (Alcohol Use Disorder) patients: A face-to-face interview and a telephone interview at treatment initiation (M0) and 6 months after programme initiation (M6)
  Administration of socio-economic questionnaires and a Brief Evaluation of Alcohol-Related Neuropsychological Impairment (BEARNI) before, and 6 months after inclusion in the therapeutic education programme.

INTERVENTIONS:
Behavioral: "Choizitaconso" - therapeutic patient education programme — Choizitaconso is a therapeutic patient education programme that teaches psychosocial skills to people with alcohol use disorder (PWAUD), to help them (re)establish controlled drinking and reduce harms.
  It lasts for 10 weeks for each participant and consists of the following 5 modules, including one optional module focusing on the family environment:
  1. Understand the mechanisms that trigger and/or maintain alcohol-related difficulties
  2. Plan and evaluate personalized controlled drinking strategies
  3. Understand and identify external and internal influences (e.g., thoughts and emotions), identify and manage risk situations
  4. Identify alcohol effects and alcohol-related expectations (by developing self-observation skills)
  5. Family environment: learning how to evaluate and take care of oneself (e.g., how to express feelings)
  Each module consists of 2 to 4 collective workshops that each last 120 minutes and involve 5 to 10 persons.
  Groups: Former therapeutic education participants; Intervention group (current therapeutic education participants)

SUMMARY:
Alcohol is the most harmful psychoactive substance in terms of overall damage. Although abstinence remains the objective of most pharmacological and non-pharmacological approaches addressing alcohol use disorder (AUD), new therapeutic objectives of reduced alcohol intake and controlled-drinking have emerged.

ETHER ("Education THEérapeutique pour la Réduction des dommages en alcoologie" or therapeutic education for the reduction of alcohol-related harms) is an ongoing, multicentre, community-based mixed-methods study, which aims to evaluate the innovative therapeutic patient education (TPE) programme named "Choizitaconso". This programme teaches psychosocial skills to people with alcohol use disorder (PWAUD), to help them (re)establish controlled drinking and reduce harms.

The evaluation of the programme will rely on a sequential explanatory design, where the qualitative study (16 semi-structured interviews) will assist in explaining and interpreting the findings of the controlled before-and-after quantitative study.

DETAILED DESCRIPTION:
ETHER's quantitative component is a 6-month controlled study which evaluates the effectiveness of "Choizitaconso" by comparing 30 PWAUD following the programme with a control group of 60 PWAUD not following it. All 90 PWAUD are individually interviewed using standardized face-to-face and phone-based interviews.

34 questions on alcohol-related harms were identified in the international literature and approved by the PWAUD community. The sum of these harms, considered as a measure of the individual "burden" related to alcohol use, will be used as principal outcome.

Secondary outcomes are quantity and frequency of alcohol consumption, craving for alcohol, coping strategies, Health-Related Quality of Life (HRQL), self-confidence to resist drinking, anticipated and internalized stigma, treatment self-regulation, anxiety and depressive symptoms, alcohol-related neuropsychological impairments and capabilities (i.e., a measure of wellbeing for the general adult population, used in economic evaluations).

Primary and secondary outcomes will be collected in face-to-face and phone-based interviews at enrolment and 6 months after enrolment. We will use a binomial test and linear regression models to assess the impact of the TPE programme on changes in the principal and secondary outcomes, while adjusting for other correlates and confounders.

The study's qualitative component comprises semi-structured interviews of 16 PWAUD who completed the TPE programme at least 6 months before the interview. Qualitative interviews will be analysed using thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* fluent in French speaker
* able to provide written, informed consent
* reachable by phone
* followed-up for Alcohol Use Disorder

Exclusion Criteria:

* cocaine or opiate dependence
* being a legally-protected adult (tutorship, curatorship)
* being pregnant
* participation in another study during the duration of follow-up (6 months)
* having severe cognitive impairment which could conflict with successful group work

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consist in adults with alcohol use disorder eligible to participate to a therapeutic patient education programme.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Community-validated alcohol-related harms | Compared after 6 months between the intervention- and the control group.
  We selected as principal outcome the number of experienced alcohol-related harms (ranging between 0 and 34) as a measure of the individual alcohol-related "burden".
  34 questions on alcohol-related harms (physical, social and behavioural consequences) were identified by and with the community of PWAUD during several working sessions.
  Alcohol-related harms assessment is scheduled at enrolment (i.e., before the TPE programme initiation for the intervention group) and 6 months later.

SECONDARY OUTCOMES:
Health-related Quality of life (SF-12v2 health survey) | Compared after 6 months between the intervention- and the control group.
  A validated measure of physical and mental
Average alcohol consumption (AUDIT-C) | Compared after 6 months between the intervention- and the control group.
  Frequency and quantity of alcohol use
Craving | Compared after 6 months between the intervention- and the control group.
  Self-reported control over alcohol consumption, and feelings related to alcohol (5 questions)
Stigma | Compared after 6 months between the intervention- and the control group.
  11 questions on anticipated and internalized stigma drawn from the Substance Use Stigma Mechanism Scale (SU-SMS)
Anxiety and depressive symptoms (HAD) | Compared after 6 months between the intervention- and the control group.
  HAD anxiety and depressive symptoms scale
Alcohol-Related Neuropsychological Impairments (BEARNI) | Compared after 6 months in the intervention group
  The Brief Evaluation of Alcohol-Related Neuropsychological Impairment (BEARNI) test is a clinical screening tool, assessing verbal episodic memory, visuospatial abilities, working memory, executive functioning
Coping strategies (Brief COPE) | Compared after 6 months between the intervention- and the control group.
  28 questions on cognitive and behavioural efforts to cope with stress in everyday life (trait coping)
Capability (ICECAP-A questionnaire) | Compared after 6 months between the intervention- and the control group.
  A measure of wellbeing for the general adult population, used in economic evaluations.
  5 questions on attachment, stability, achievement, enjoyment and autonomy
Treatment self-regulation | Compared after 6 months between the intervention- and the control group.
  Reasons for entering treatment or engaging in healthy behaviour Adaptation of the "Treatment Questionnaire Concerning Diabetes" including 2 subscales: autonomous regulation and controlled regulation
Self-confidence to resist drinking (Brief Situational Confidence Questionnaire) | Compared after 6 months between the intervention- and the control group.
  Confidence to resist (or control) drinking in high-risk situations

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CSAPA Convergence, Avignon
  - ANPAA 04, Digne-les-Bains
  - Clinique Saint Barnabé, Marseille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barre T, Ramier C, Antwerpes S, Costa M, Bureau M, Maradan G, Di Beo V, Cutarella C, Leloutre J, Riccobono-Soulier O, Hedoire S, Frot E, Vernier F, Vassas-Goyard S, Dufort S, Protopopescu C, Marcellin F, Casanova D, Coste M, Carrieri P. A novel community-based therapeutic education program for reducing alcohol-related harms and stigma in people with alcohol use disorders: A quasi-experimental study (ETHER study). Drug Alcohol Rev. 2023 Mar;42(3):664-679. doi: 10.1111/dar.13605. Epub 2023 Jan 31. PMID 36721903
- [Result] Antwerpes S, Costa M, Coste M, Bureau M, Maradan G, Cutarella C, Leloutre J, Riccobono-Soulier O, Hedoire S, Frot E, Vernier F, Vassas-Goyard S, Barre T, Casanova D, Carrieri P. Evaluation of a novel therapeutic education programme for people with alcohol use disorder in France: a mixed-methods intervention study protocol (ETHER). Harm Reduct J. 2022 Jan 10;19(1):2. doi: 10.1186/s12954-021-00587-0. PMID 35012570